CLINICAL TRIAL: NCT00337064
Title: Phase I/II Trial to Evaluate Partial Breast Radiation to the Region of the Lumpectomy Cavity Using Intensity Modulated Radiation in Elderly Women With Breast Cancer
Brief Title: Partial Breast Radiation to the Lumpectomy Cavity With IMRT in Elderly Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC0601
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2006-06-15 (Estimated); Status verified 2006-05

CONDITIONS: Stage I Breast Cancer
Keywords: Breast cancer treatment; Partial breast radiation; Radiation Therapy; Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: Radiation Therapy

SUMMARY:
The standard treatment for women with invasive breast cancer is local excision follow by whole breast radiation. The local recurrence rates are low, side effects are low, and the cosmetic outcome is excellent. The treatments, however, need to be given daily for 5 1/2 to 6 1/2 weeks, making the treatment difficult, particularly for the elderly and for women who need to travel long distances for the therapy. The goal of this study is to determine the toxicity and efficacy of giving the radiation in a shorter time, using higher daily doses of radiation.

The risk of recurrence in the elderly population is lower, and since majority of recurrences occur close to the area where the tumor previously was, it is hypothesized that radiation to that area of the breast would be sufficient to obtain low risk of recurrence. When a smaller volume of tissue is treated, more radiation can be given daily, and therefore the treatment can be shortened. The risk of side effects increases as the dose per daily treatment increases. Therefore, the goal is to study the short term side effects, long term side effects, and cosmetic outcome of daily radiation using higher daily doses for shorter period of time. We will also follow the recurrence rate. Because less of the breast tissue will be treated, there may be a small increased risk of recurrence. Because the higher fraction size can result in more side effects we will be using intensity modulated radiation (IMRT). IMRT is the most advanced individually tailored radiation treatment technique that results in the least amount of side effects. It allows tight monitoring of the dose in the untreated breast.

Seventy five women diagnosed with stage I breast cancer will participate. Participants must have a lumpectomy, clear margins and no lymphovascular invasion to be eligible. A treatment planning CT scan will be obtained. If the lumpectomy cavity can be clearly delineated, an IMRT plan will be generated with predefined strict dose requirement criteria. The patients will be treated once daily, 5 days a week, for a total of 10 treatments (instead of standard 28-33). The patients will be evaluated for toxicity weekly during the treatment, and weekly for additional 4 weeks. At each of these evaluations, they will fill out a short 10 minute questionnaire detailing their side effects. Follow-up will continue every 3 months for 3 years, and every 6 months for 2 more years. At each of these follow-ups a short questionnaire will be filled out by the patients detailing any toxicity, as well as their perception of the cosmetic outcome. A cosmesis questionnaire will be also be filled out by the evaluating physician before radiation, at 6, 12, 18, and 24 months, and yearly for 3 more years. A total of 5 years of follow-up is planned. Participants will also have the option of consenting to the photograph portion of the study. Those who do will have photographs taken of their breasts (excluding faces) at the time they complete the cosmetic questionnaire, to evaluate the cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Stage I ductal breast cancer,
* Status post lumpectomy/partial mastectomy and axillary dissection or sentinel lymph node biopsy
* Age over 65
* Pathologically negative margins
* No lymphovascular invasion
* Able to begin radiation treatment 3-8 weeks post surgery, unless receiving chemotherapy first
* Lumpectomy cavity is visible in CT
* Patient is female

Exclusion Criteria:

* Lymphovascular invasion
* Positive nodes or tumor size greater than 2 cm
* Positive margins
* Age less than 65
* Patient is male

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75
Dates: Start 2006-06

PRIMARY OUTCOMES:
Acute sdie effects
Percent of times that the target definition on planning CT is attained
Percent of times that the treatment is within the prescription goals

SECONDARY OUTCOMES:
Set up variations
Subacute and long-term side effects
Cosmetic outcome
Percent experiencing local failure, time to recurrence and percent who can be retreated with radiation following recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Heimann, M.D., Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care, Radiation Oncology, Burlington, Vermont, United States